CLINICAL TRIAL: NCT07290712
Title: Post-Intensive Care Syndrome - Multicentre Prospective Registry Database of the DACH Region
Acronym: PICS-DACH
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Wuerzburg (Other); University Hospital Augsburg (Other)
Responsible Party: Principal Investigator, Stefan Schaller, Professor of Anaesthesia and Anaesthesiological Intensive Care Medicine, Medical University of Vienna
Other Study IDs: PICS-DACH
Record Dates: First submitted 2025-09-29; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: PICS; PICS-F
Keywords: PICS; PICS-F; ICU; Intensive Care Unit; Critical Care; Critical Illness; Post Intensive Care Syndrome; Post Intensive Care Syndrome Family
MeSH Terms: conditions — Critical Illness; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — A blood sample may be collected by centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-Intensive Care Syndrome (PICS) refers to long-term cognitive, physical, and psychological impairments that can arise after intensive care treatment. These symptoms may begin within 24 hours of ICU admission and persist for years. Affected patients and their families (PICS-F) face significant burdens, with up to 94% of relatives impacted. Given its high prevalence and socioeconomic impact, this prospective registry study aims to identify risk factors and long-term consequences of PICS and PICS-F.

The study consists of six modules, starting with data collection during ICU stays and continuing with follow-ups at various intervals post-discharge (up to five years). The primary goal is to investigate diagnostic and therapeutic strategies, while secondary objectives include identifying risk factors, determining impairment severity, and exploring biological mechanisms. Standardized questionnaires and biological samples (blood) are used for data collection.

DETAILED DESCRIPTION:
BACKGROUND Post-Intensive Care Syndrome (PICS) refers to newly occurring or intensified cognitive, physical, and psychological long-term effects, as well as pain and socioeconomic effects resulting from intensive care treatment. Symptoms can appear as early as 24 hours after admission to the intensive care unit (ICU) and persist for 5-15 years after discharge. The rate of affected individuals is very high. Three months after discharge due to an illness requiring intensive care, 64% of survivors were impaired in at least one of the three functional areas, and 56% were impaired after 12 months. The hospitalization of a close relative in the ICU affects the entire family system, i.e., all people with whom the patients have a significant relationship. The effects on the family or relatives are referred to as Post-Intensive Care Syndrome-Family (PICS-F), which represents a significant burden for up to 94% of relatives. PICS and PICS-F are therefore of high socioeconomic importance.

RELEVANCE Given the significant impact of PICS on patients, their families, and the socioeconomic system, gaining insights into the prevalence of risk factors and PICS criteria during ICU stay, as well as PICS and PICS-F after ICU discharge and hospital release, is highly valuable.

DESIGN

The study is divided into the following six modules:

1. ICU module
2. Post-ICU module 2: a) 1-3 months + 6 months, b) 1, 2, 5 years
3. Environment module
4. Psychiatry module
5. Translational module
6. Family system module (PICS-F) The participating centers take part in at least the first module, the ICU module, in which the risk factors and PICS as well as PICS-F domains are recorded during the intensive care stay. Depending on local conditions, capacity, and resources, the participating centers optionally participate in modules 2 to 6. In the individual modules, there is also the option of participating in a mode available to all centers or specialized for individual centers (e.g., functional tests that can only be performed in a PICS outpatient clinic (PICA)). For centers without PICA, follow-up observation is carried out, for example, via questionnaires. The corresponding mode of participation with and without PICA is displayed accordingly in the individual modules.

PRIMARY OBJECTIVE

• The primary objective of the prospective registry is to record and investigate the risk factors, diagnostic and therapeutic options for PICS and PICS-F.

SECONDARY OBJECTIVES

* Recording the frequency of multiple risk factors for and the manifestation of PICS and PICS-F during and after treatment in an intensive care unit.
* Recording the rate of risk factors, especially the modifiable risk factors of PICS in different disease entities, such as sepsis, delirium, and other underlying diseases requiring intensive care.
* Determination of cut-off values and rates of significant cognitive, physical and psychological impairments as well as pain.
* Assessment of the significance for PICS between and within individual dimensions of PICS.
* Estimation of incidence based on risk factors or different cut-off values for scores to define significant limitations at the cognitive, physical and psychological levels as well as chronic pain.
* Determination and investigation of the influence of relevant external and internal environmental factors that contribute to the development and course of PICS/PICS-F.
* Identification of molecular biological or pathophysiological processes of PICS.

PROCEDURE

1. Examination using standardized questionnaires during intensive care. The aim is to record cognitive, physical, and psychological functional impairments as well as pain (= PICS and PICS-F rates) while still in the intensive care unit. The patient and their relatives and friends are interviewed.
2. Follow-up examination using standardized questionnaires in the PICS outpatient clinic 1-3 and 6 months after discharge from the intensive care unit. The aim of these appointments is to record cognitive, physical, and psychological functional impairments as well as pain.
3. Completion of standardized questionnaires to record cognitive, physical, and psychological functional impairments as well as pain (1, 2, and 5 years after discharge from the intensive care unit; this can be done by telephone, electronically, by mail, via telemedicine, or in PICA).
4. Blood samples for the creation of a biobank (depending on follow-up appointments at the PICS study outpatient clinic: 4-7x 27ml each; timing: during ICU (inclusion (> 72h ICU stay) and ICU discharge), 1-3 months, 6 months and, if applicable, 1, 2, and 5 years after ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ICU stay longer than 72 hours will be included

Exclusion Criteria:

* Age < 18 years old
* Patients who receive end-of-life care at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Post-Intensive Care Syndrome (PICS) | up to 5 years
  Frequency of PICS diagnosis defined as the presence of at least one new or worsened impairment in one of the PICS domains (number/percentage)

SECONDARY OUTCOMES:
Frequency of PICS sub-domains | up to 5 years
  Frequency of diagnosis of PICS-subdomains
Frailty status | up to 5 years
  Frailty status assessed by the Clinical Frailty Scale (CFS; score 1-9, higher scores indicate worse frailty).
Post-Intensive Care Syndrome symptoms assessed by the PICS Questionnaire (PICSq) | up to 5 years
  PICS symptoms assessed by the PICSq (validated questionnaire 0-45 points; higher scores indicate greater impairment).
Physical function assessed by the Barthel Index | up to 5 years
  Change in activities of daily living, assessed by the Barthel Index (score 0-100; higher scores indicate better function).
Physical function assessed by the Timed Up-and-Go Test | up to 5 years
  Change in mobility, assessed by the Timed Up-and-Go(time in seconds; longer times indicate worse performance).
Physical function assessed by Handgrip Strength | up to 5 years
  Muscle strength, assessed by handgrip dynamometry (maximum grip strength in kg; higher values indicate better function).
Physical function assessed by the 6-Minute Walk Test (6MWT) | up to 5 years
  6MWT (distance walked in meters; higher values indicate better function).
Physical function assessed by the 2-Minute Walk Test (2MWT) | up to 5 years
  ´2MWT (distance walked in meters; higher values indicate better function).
Physical function assessed by the SPPB | up to 5 years
  Physical function, assessed by the Short Physical Performance Battery (SPPB, score 0-12; higher scores indicate better performance).
Nutritional status assessed by the MNA | up to 5 years
  Nutritional status, assessed by the Mini Nutritional Assessment (MNA, score 0-30; higher scores indicate better nutritional status).
Health-related quality of life assessed by EQ-5D-5L | up to 5 years
  Health-related quality of life, assessed by the EQ-5D-5L (index score; higher values indicate better quality of life).
Disability assessed by the WHO Disability Assessment Schedule (WHODAS 2.0) | up to 5 years
  Disability, assessed by the WHODAS 2.0, with higher scores indicating greater disability.
Cognitive function assessed by the MiniCog | up to 5 years
  Cognitive function, assessed by the MiniCog (score 0-5; higher scores indicate better cognition).
Cognitive function assessed by the Animal Naming Test | up to 5 years
  Verbal fluency, assessed by the Animal Naming Test (number of animals named in 60 seconds; higher values indicate better cognition).
Cognitive function assessed by the RBANS | up to 5 years
  Cognition, assessed by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS; higher scores indicate better cognition).
Cognitive function assessed by the TMT | up to 5 years
  Executive function, assessed by the Trail Making Test (TMT A and B, completion time in seconds; longer times indicate worse performance).
Depression assessed by the PHQ | up to 5 years
  Depression severity, assessed by the Patient Health Questionnaire (PHQ, higher scores indicate worse depression).
Anxiety assessed by the GAD | up to 5 years
  Anxiety severity, assessed by the Generalized Anxiety Disorder scale (GAD, higher scores indicate worse anxiety).
PTSD symptoms assessed by the IES-R | up to 5 years
  Post-traumatic stress disorder (PTSD) symptoms, assessed by the Impact of Event Scale - Revised (IES-R; higher scores indicate worse PTSD symptoms).
Pain assessed by the McGill Pain Questionnaire | up to 5 years
  Pain severity, assessed by the McGill Pain Questionnaire (higher scores indicate worse pain).
Frequency of dysphagia | up to 5 years
  Frequency of clinically diagnosed swallowing disorder (number / percentage)
Work ability and disability days | 5 years
  Change in employment status and number of disability days from baseline to 5 years, assessed by self-report (more disability days indicate worse outcome).
Psychiatric or psychotherapeutic care utilization | 5 years
  Use of psychiatric or psychotherapeutic services (yes/no), assessed from baseline to 5 years.
Noise annoyance assessed by the 11-point numeric noise-annoyance scale | 5 years
  Change in noise annoyance from baseline to 5 years, assessed by the 11-point numeric scale (0-10; higher scores indicate higher annoyance).
Noise annoyance assessed by the 5-point verbal scale | 5 years
  Change in noise annoyance from baseline to 5 years, assessed by the 5-point verbal scale (1-5; higher scores indicate higher annoyance).
Noise sensitivity assessed by the LEF-K questionnaire | 5 years
  Change in noise sensitivity from baseline to 5 years, assessed by the LEF-K (higher scores indicate greater sensitivity).
ICU environmental exposure measured by HIAwear/Sensorbox | 5 years
  Change in ICU environmental exposure from baseline to 5 years, measured continuously with HIAwear/Sensorbox (parameters include noise, light, particulate matter, temperature, humidity; higher values indicate greater exposure).
Atmospheric environmental exposure (ozone, nitrogen oxides, carbon monoxide, particulate matter) | 5 years
  Change in atmospheric exposure from baseline to 5 years, assessed by pollutant concentrations (O3, NO, NO2, NOx, CO, PM1, PM2.5, PM10; higher values indicate greater exposure).
Anxiety and depression in relatives assessed by the HADS | 5 years
  Change in anxiety and depression symptoms of relatives from baseline to 5 years, assessed by the HADS (score 0-21; higher scores indicate worse symptoms).
Post-traumatic stress in relatives assessed by the IES-R | 5 years
  Change in PTSD symptoms of relatives from baseline to 5 years, assessed by the IES-R (higher scores indicate worse PTSD symptoms).
Work ability of relatives | 5 years
  Change in work status and disability days of relatives from baseline to 5 years, assessed by self-report (more disability days indicate worse outcome).
Psychiatric or psychotherapeutic care utilization by relatives | 5 years
  Use of psychiatric or psychotherapeutic services (yes/no), assessed in relatives from baseline to 5 years.
Body resistance (R) | up to 5 years
  Body resistance (R) measured by BIA (Body impedance analysis)
Body reactance (Xc) | up to 5 years
  Body reactance (Xc) measured by BIA (Body impedance analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Medical University of Vieanna; Bjoern Weiss, MD, Principal Investigator — Charite University, Berlin, Germany; Claudia Denke, Dr., Principal Investigator — Charite University, Berlin, Germany; Patrick Meybohm, MD, Principal Investigator — Wuerzburg University Hospital; Philipp Simon, MD, Principal Investigator — Universitätsklinikum Augsburg; Claudia Spies, MD, Principal Investigator — Charite University, Berlin, Germany; Christian Stoppe, MD, Principal Investigator — Wuerzburg University Hospital; Manfred Weiss, MD, Principal Investigator — Universitätsklinikum Augsburg; Marion Wiegele, MD, Principal Investigator — Medical University of Vienna
Locations (4):
- Medical University of Vienna, Vienna, Vienna, Austria
- Germany (3):
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: The Study Protocol will be public. IPD can only be shared in a research collaboration with other researchers if data protection regulations allow it and after signing a data sharing and research collaboration contract. Start date after publication of the first PICS-DACH data.
Access Criteria: The Study Protocol will be public. IPD can only be shared in a research collaboration with other researchers if data protection regulations allow it and after signing a data sharing and research collaboration contract.
URL: https://www.pics-dach.eu

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Jeong YJ, Kang J. Development and validation of a questionnaire to measure post-intensive care syndrome. Intensive Crit Care Nurs. 2019 Dec;55:102756. doi: 10.1016/j.iccn.2019.102756. Epub 2019 Sep 12. PMID 31522829
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- See also: Webpage of the PICS-DACH Consortium — https://www.pics-dach.eu